CLINICAL TRIAL: NCT07191249
Title: A Phase 2, Multicenter, Open-Label Trial to Evaluate Efficacy and Safety of Subcutaneous (SC) Mosunetuzumab in Previously Untreated Low Tumor Burden Follicular Lymphoma (LTB-FL).
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0691-24-TLV
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma
Keywords: Fullicular Lymphoma; Mosunetuzumab
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, single-arm, open-label study evaluating the efficacy and safety of subcutaneous Mosunetuzumab in patients with low tumor burden follicular lymphoma. All participants receive the same intervention without randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with follicular lymphoma with low tumor burden who have not been previously treated (Experimental): In this study, Mosunetuzumab will be administered subcutaneously over 8 treatment cycles: 5 mg on Day 1 of Cycle 1, followed by 45 mg in all subsequent cycles.
  Interventions: Drug: Mosunetuzumab is a bispecific monoclonal antibody targeting CD20 on B cells and CD3 on T cells, redirecting T cells to eliminate malignant B cells.

INTERVENTIONS:
Drug: Mosunetuzumab is a bispecific monoclonal antibody targeting CD20 on B cells and CD3 on T cells, redirecting T cells to eliminate malignant B cells. — In this study, Mosunetuzumab will be administered subcutaneously over 8 treatment cycles: 5 mg on Day 1 of Cycle 1, followed by 45 mg in all subsequent cycles.

SUMMARY:
This is a multi-center, open-label, interventional clinical trial designed to evaluate the efficacy and safety of subcutaneous (SC) Mosunetuzumab as a first-line immunotherapy in patients with low tumor burden follicular lymphoma (LTB-FL), defined by the absence of GELF criteria.

Eligible patients will undergo screening and, upon signing an Informed Consent Form, will receive their first dose of SC Mosunetuzumab.

Mosunetuzumab is administered via SC injection without the need for mandatory hospitalization. The first cycle lasts 21 days, followed by subsequent 28-day cycles. In Cycle 1, Mosunetuzumab is given on Day 1 (5 mg), Day 8 (45 mg), and Day 15 (45 mg). From Cycle 2 onward, a single 45 mg dose is administered on Day 1 of each cycle. Treatment continues for up to 8 cycles (approximately 6 months).

Patients will be monitored for disease status according to standard clinical practice. After completing active treatment, they will enter a post-treatment follow-up phase. Premedication with dexamethasone (20 mg) is mandatory in Cycle 1 and optional in later cycles. Acetaminophen and diphenhydramine may also be administered.

All patients will continue study treatment as per the Schedule of Activities or until premature discontinuation. After treatment discontinuation, disease status assessments will occur approximately every 3 months for up to 24 months. During post-treatment follow-up, PET-CT scans for disease evaluation will be performed every 6 months, as applicable. Patients not under active follow-up will be contacted annually to collect data on disease status and survival.

Throughout the trial, the following data will be collected (as applicable): demographics and baseline characteristics (including sex, age, race, height, and weight), medical history, details of initial diagnosis and treatment history, concomitant medications, adverse events (AEs), serious adverse events (SAEs), disease response, and survival status.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Histologically confirmed classic FL (cFL) (according to WHO-HEAM4R classification)
* Low tumor burden by GELF criteria
* No prior therapy except surgery or radiotherapy for disease that was previously localized
* Ann Arbor Stage III or IV disease
* Bi-dimensionally measurable FDG-avid disease defined by at least one single node or tumor lesion > 1.5 cm assessed by CT scan and/or clinical examination
* Adequate hematologic function defined as follows without growth factors or blood product transfusion within 14 days of first dose of study drug administration:

  1. Hemoglobin, without transfusion, 9 g/dL
  2. ANC 1.0 109/L
  3. Platelet count 75 109/L;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Patient can understand and sign the Informed Consent Form (ICF), can communicate with the Investigator, can understand and comply with the requirements of the protocol

Exclusion Criteria:

* 1. An active viral infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) defined by detectable viral DNA in the blood by PCR. Patients with HIV are eligible provided an undetectable viral load and a CD4 count > 200 cell/mcl
* 2. Any of the following laboratory abnormalities:

  1. Total Bilirubin or GGT or AST or ALT > 3 X ULN.
  2. Creatinine Clearance calculated by Cockcroft and Gault Formula < 40 ml/min
* Presence or history of CNS involvement by lymphoma
* 4. Prior history of malignancies other than Lymphoma (except for Basal Cell or Squamous Cell Carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 2 years
* Contraindication to use Mosunetuzumabor known sensitivity or allergy
* Pregnant or lactating females
* 7. Female patients of childbearing potential who cannot or do not wish to use an effective method of contraception, during the study treatment and for 3 months thereafter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Overall response rate (ORR) at the end of treatment (6 months) using the Lugano criteria | 6 months
  It refers to the proportion of patients who experience a predefined reduction in tumor size as a result of treatment.

SECONDARY OUTCOMES:
1. Incidence of adverse events (AEs) and abnormal laboratory test results from first dose through 90 days after administration of last dose; | through 90 days after administration of last dose;
Progression free survival (PFS), complete metabolic response rate (CRR), duration of response (DOR), duration of complete response, time to next systemic anti-lymphoma treatment (TTNT) and overall survival (OS) at 12 and 24 months | at 12 and 24 months
Patient reported outcomes (PROs) according to the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) subscale. | 6 months (after last drug administration

OTHER OUTCOMES:
Exploratory Biomarker Research Endpoints: Longitudinal measurement of ctDNA in the peripheral blood (PB), before and during treatment, at disease progression, at CR and one year after achievement of CR, as a biomarker for long-term remission | one year after achievement of CR, a
Evaluating the treatment-induced dynamics and molecular signatures of the non-tumor lymphocytic and myeloid compartments, performing consecutive flow cytometry, single cell RNA sequencing (scRNA-seq) and epigenetic studies, and correlation with outcome; | one year after achievement of CR
  Time points: before and during treatment, at disease progression, at CR and one year after achievement of CR.
Analyzing tumor microenvironment (TME) in lymph nodes pre-treatment at disease progression, at CR and one year after achievement of CR by performing scRNA-seq; | one year after achievement of CR
Evaluating the association between patient's microbiome and response to treatment | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Irit Avivi, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center